CLINICAL TRIAL: NCT05037357
Title: Verification of Harmonization of Plasma Epstein-Barr Virus DNA Measurements at Multiple Centers in NPC Epidemic Regions
Brief Title: Verification of Harmonization of Plasma Epstein-Barr Virus DNA Measurements
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Wuzhou Red Cross Hospital (Other); Zhongshan People's Hospital, Guangdong, China (Other)
Responsible Party: Principal Investigator, Ming-Yuan Chen, professor & chief physician, Sun Yat-sen University
Other Study IDs: SYSUCC-CMY-2021-EBV
Record Dates: First submitted 2021-08-10; First posted 2021-09-08 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal Carcinoma; plasma EBV DNA; Harmonization
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood will be collected into ethylenediaminetetraacetic acid (EDTA)-coated tubes and centrifuged, the plasma will be recovered and frozen at -80℃ until the test.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- nasopharyngeal carcinoma patients: Plasma EBV DNA quantification by quantitative polymerase chain reaction (qPCR) assays in different medical centers.
  Interventions: Diagnostic Test: Plasma EBV DNA qPCR test

INTERVENTIONS:
Diagnostic Test: Plasma EBV DNA qPCR test — Peripheral blood will be collected from each subject into an EDTA tube for the isolation of plasma.

SUMMARY:
Plasma Epstein-Barr virus (EBV) DNA will be measured in native plasma samples of nasopharyngeal carcinoma (NPC) patients, respectively, by three medical centers and a qualified laboratory in Southern China, the highest endemic area of NPC. Passing-Bablok regression and difference plots will be used to compare results from each center to the all-method median and mean values. Agreement among methods will be evaluated against bias derived from a biological variation.

DETAILED DESCRIPTION:
The investigators intend to collect EBV DNA positive plasma samples of NPC patients, distribute the samples to four test centers and compare the measurement results to obtain the current status of the agreement of plasma EBV DNA measuring at different centers with various measurement systems in the endemic regions of NPC. A series of statistical analyses including Cohen's Kappa, intraclass correlation coefficient, and Passing-Bablok regression will be adopted for the consistency test. A harmonization study by using the same calibrators will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-70 years
* Histologically confirmed NPC or Non-NPC with positive plasma cell-free EBV DNA

Exclusion Criteria:

* unsatisfactory performance status: Karnofsky scale (KPS) <= 70
* Any severe intercurrent disease
* Any contraindication of blood sampling

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: NPC patients or Plasma EBV DNA positive people
Sampling Method: Non-Probability Sample
Enrollment: 370 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Plasma EBV DNA | 1 Day
  copy number of EBV DNA in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Yuan Chen, MD, PhD, Study Chair — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided